CLINICAL TRIAL: NCT00103597
Title: Efficacy of Therapeutic Interventions for Orthostatic Hypotension in Parkinson's Disease and Multiple System Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Royal Brisbane and Women's Hospital (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2004/135; 2004/135
Record Dates: First submitted 2005-02-11; First posted 2005-02-14 (Estimated); Last update posted 2005-10-20 (Estimated); Status verified 2005-07

CONDITIONS: Parkinson's Disease; Multiple System Atrophy; Orthostatic Hypotension
Keywords: Orthostatic hypotension; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Hypotension, Orthostatic | interventions — Fludrocortisone; Domperidone

INTERVENTIONS:
Drug: Fludrocortisone
Drug: Domperidone
Behavioral: Conservative Measures for Orthostatic Hypotension

SUMMARY:
Patients with Parkinson's Disease or Multiple System Atrophy (MSA), and symptoms of orthostatic hypotension, are eligible for the study. Each patient will have three weeks of conservative therapy, three weeks of therapy with fludrocortisone, and three weeks of therapy with domperidone. Autonomic testing, a symptom questionnaire, bedside blood pressure testing, and Unified Parkinson Disease Rating Scale (UPDRS) will be performed after each intervention.

DETAILED DESCRIPTION:
Enrolled patients, ages 40-95, must have Parkinson's or MSA, diagnosed by a neurologist, and symptoms of orthostatic hypotension. Each patient will fill out two validated questionnaires to determine if they are candidates for the study. Baseline patient details, such as their medications and UPDRS, will be recorded. Medications must be held stable during the period of the study.

Each patient will then have three weeks of conservative therapy, three weeks of therapy with fludrocortisone, and three weeks of therapy with domperidone. Autonomic testing, a symptom questionnaire, bedside blood pressure testing, and UPDRS will be performed after each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients residing in Queensland Australia
* Age 40-95
* Parkinson's Disease or MSA diagnosed by a neurologist
* Symptoms of orthostatic hypotension, as defined by 2 validated questionnaires

Exclusion Criteria:

* Patients with acute cardiomyopathy or cardiac condition
* Patients unable to give consent
* Patients not stable on their Parkinsonian medications
* Patients with another cause for autonomic neuropathy

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-01; Study Completion 2005-09

PRIMARY OUTCOMES:
Efficacy of conservative treatment, domperidone, and fludrocortisone for patient's subjective symptoms of orthostatic hypotension, and on objective autonomic testing

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Schoffer, MBBS, Principal Investigator — Movement Disorders Fellow
Locations (1):
- Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Veazie S, Peterson K, Ansari Y, Chung KA, Gibbons CH, Raj SR, Helfand M. Fludrocortisone for orthostatic hypotension. Cochrane Database Syst Rev. 2021 May 17;5(5):CD012868. doi: 10.1002/14651858.CD012868.pub2. PMID 34000076